CLINICAL TRIAL: NCT03454022
Title: Decision-Aid for Renal Therapy Pilot Trial (DART Pilot Trial)
Brief Title: Decision-Aid for Renal Therapy Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Tufts Medical Center (Other); Saint Elizabeth's Medical Center (Unknown)
Responsible Party: Principal Investigator, Keren Ladin, Assistant Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12345
Record Dates: First submitted 2018-01-16; First posted 2018-03-05 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Renal Insufficiency, Chronic; Kidney Failure, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Participants (patient-caregiver dyads) will be randomized to receive either usual care education (a pamphlet published by the National Kidney Foundation, "Choosing a Treatment for Kidney Failure," or usual care education plus DART.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Participants receive an educational pamphlet from the National Kidney Foundation, "Choosing a Treatment for Kidney Failure."
  Interventions: Behavioral: Choosing a Treatment for Kidney Failure
- DART (Experimental): Participants receive an educational pamphlet from the National Kidney Foundation, "Choosing a Treatment for Kidney Failure." They also receive a link to access the web-based decision-aid program, Decision-Aid for Renal Therapy (DART). Participants may access this program using a computer at home throughout the duration of the trial. Those who do not have a computer with web access at home are assisted in watching the program in the clinic.
  Interventions: Behavioral: DART; Behavioral: Choosing a Treatment for Kidney Failure

INTERVENTIONS:
Behavioral: DART — A one-hour long web-based decision-aid program that explains treatment options for end-stage renal disease, including the benefits and risks of each treatment option.
  Arms: DART
Behavioral: Choosing a Treatment for Kidney Failure — This is an educational pamphlet published by the National Kidney Foundation.

SUMMARY:
Successful communication between patients, caregivers, and physicians can improve how patients feel about their treatment. Our recent studies of older dialysis patients find, however, that many patients do not engage in this type of communication about treatment options. This study aims to determine whether the Decision-Aid for Renal Therapy (DART), a web-based program, can improve shared decision-making (decisions where patients are actively engaged) among patients, caregivers, and physicians, and improve certainty and satisfaction in treatment decisions.

DETAILED DESCRIPTION:
Successful end-of-life communication between patients, caregivers, and physicians is associated with superior psychosocial outcomes, less intensive treatment, greater satisfaction, and higher likelihood of death at home. The Decision-Aid for Renal Therapy (DART) is an interactive web-based decision-aid that can empower patients and caregivers to select the treatment choice for chronic kidney disease that best suits them. DART was developed using a rigorous, validated, patient-engaged process and helps clarify decision-points and tradeoffs by providing individualized information about outcomes that matter most to patients. DART is designed to promote shared decision-making between patients, caregivers, and physicians and align preferences with treatment received.

Although proven effective and in current use in the general population, DART's effectiveness in an older population is unclear. The purpose of this project is to conduct a pilot study of DART's feasibility and effectiveness to improve end-of-life planning and shared decision-making among older end-stage renal disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stages 4 or 5, not currently on dialysis
* Age >=70
* English-speaking
* Willingness to be randomized to DART
* Able to sign informed consent
* 5-year kidney failure risk probability > 15% using [www.kidneyfailurerisk.com]
* Glomerular filtration rate (GFR) < 30

Exclusion Criteria:

* Non-English speaking

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Completion of advance directives at 3 months. | Assessed at 3 months
  Participants will be asked if they have completed an advance directive.
Change in baseline Decisional Conflict Scale score at 3 months. | Assessed in patients at 3 months.
  Measures personal perceptions of: a) uncertainty in choosing options; b) modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and c) effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).

SECONDARY OUTCOMES:
Congruence in patient-caregiver goals of care | Assessed in patients and caregivers at 6 months.
  Patients and caregivers are each administered a questionnaire to determine what the patient's goals of care are at the end of life. The congruence (agreement) between the stated preferences of the patient and caregiver will be assessed at 6 months.
Change in baseline overall patient satisfaction score from the Canadian Health Care Evaluation Project (CANHELP) questionnaire at 3 months. | Assessed in patients at 3 months.
  A survey instrument that evaluates satisfaction with care for older patients with life threatening illnesses, and their family members. The overall CANHELP Lite satisfaction score is calculated as the unweighted average of all answered questions. The score is then rescaled to range between 0 (worst possible value) to 100 (best possible value).
Change in baseline overall caregiver satisfaction score from the Canadian Health Care Evaluation Project (CANHELP) questionnaire at 3 months. | Assessed in caregivers at 3 months.
  A survey instrument that evaluates satisfaction with care for older patients with life threatening illnesses, and their family members. The overall CANHELP Lite satisfaction score is calculated as the unweighted average of all answered questions. All scores are rescaled to range between 0 (worst possible value) to 100 (best possible value).

CONTACTS AND LOCATIONS:
Overall Officials: Keren Ladin, PhD, Principal Investigator — Tufts University
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Brighton, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (4):
  • Study Protocol (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT03454022/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03454022/SAP_001.pdf
  • Informed Consent Form: Patient ICF (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT03454022/ICF_002.pdf
  • Informed Consent Form: Caregiver ICF (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT03454022/ICF_003.pdf